CLINICAL TRIAL: NCT03385395
Title: A Randomized, Double-blind, Parallel-group, Multicenter, Pharmacokinetic Study Comparing Weekly Intravenous Administration of OctaAlpha1 (Octapharma) With a Marketed Preparation Glassia® (Kamada Ltd.) in Subjects With Alpha-1-antitrypsin Deficiency
Brief Title: Study Comparing Weekly Intravenous Administration of OctaAlpha1 With a Marketed Preparation Glassia® in Subjects With Alpha-1-antitrypsin Deficiency
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND has been closed.
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OctaAlpha1
Record Dates: First submitted 2017-12-01; First posted 2017-12-28 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OctaAlpha1 (Experimental)
  Interventions: Drug: OctaAlpha1
- Glassia® (Active Comparator)
  Interventions: Drug: Glassia

INTERVENTIONS:
Drug: OctaAlpha1 — For OctaAlpha1 the standard weekly dose of 60mg/kg will be given for 24 consecutive infusions
  Arms: OctaAlpha1
Drug: Glassia — For Glassia the standard weekly dose of 60mg/kg will be given for 24 consecutive infusions
  Arms: Glassia®

SUMMARY:
This randomized trial is being conducted to show non-inferiority of OctaAlpha1 compared to Glassia® in terms of the serum trough levels at steady state. This will be conducted in individuals with alpha-1-antitrypsin deficiency and clinical evidence of emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Any subject who needs chronic IV augmentation and maintenance therapy with A1PI because of congenital alpha-1-proteinase inhibitor (A1PI) deficiency and clinically diagnosed emphysema
* ≥18 years of age
* Individuals with A1PI serum concentration <11 µM at screening
* Following bronchodilators:

  * Initial FEV1(pred) between 25% and 75% or
  * If the initial FEV1 was greater than 75% of predicted, a diffusing capacity of the lung for carbon monoxide (DLC O) less than 70% of predicted
* Following bronchodilators: Initial forced expiratory volume/forced vital capacity (FEV1/FVC) ratio less than 70%
* Non-smoking for at least 6 months before study treatment starts
* Able to understand and provide written informed consent
* Women of reproductive age: negative result of pregnancy test (human chorionic gonadotropin [HCG]-based assay) and agreement to use adequate contraception for the duration of the trial

Exclusion Criteria:

* Any inflammatory condition or malignant tumor in the 7 days before treatment starts that according to investigator judgment might influence the metabolism of an enzyme inhibitor such as A1PI
* More than one A1PI-deficiency related exacerbation and/or hospitalization during the 3 months before study treatment starts
* Clinically significant liver or kidney disease in the preceding 6 months before study treatment starts
* Severe gas exchange abnormality (i.e., PaCO2 ≥46 mmHg)
* Known IgA deficiency with documented antibodies against IgA
* History of hypersensitivity to blood or plasma derived products, or any component of the product
* Known presence of antibodies against A1PI
* Seropositivity for HBsAg or HCV, HIV-1/2 IgG antibodies
* Administration of A1PI products in the 4 weeks before study treatment starts
* Participating in another clinical study currently or during the 3 months before study treatment starts.
* Live viral vaccination within the last month before study treatment starts
* A current life-threatening malignancy
* Emergency operation within 3 months before study treatment starts
* History of, or suspected, alcohol or drug abuse within 1 year before study treatment starts or currently on drug abuse therapy
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of OctaAlpha1 compared to Glassia® in terms of the serum trough levels at steady state | 26 weeks
  Non-inferiority of OctaAlpha1 compared to Glassia® in terms of the serum trough levels at steady state

SECONDARY OUTCOMES:
Compare PK parameters following a single dose between the two treatment groups following principles of bio-equivalence testing (AUC) | Time period including days 1 to 14 after first infusion in study
  Compare PK parameters following a single dose between the two treatment groups calculating area under the plasma concentration-time curve (AUC)-ratio: 90% confidence interval (CI) should lie within 80%-125%.
Compare PK parameters following a single dose between the two treatment groups following principles of bio-equivalence testing (Cmax) | Time period including days 1 to 14 after first infusion in study
  Compare PK parameters following a single dose between the two treatment groups calculating maximum plasma concentration (Cmax)-ratio: 90% CI should lie within 80%-125%
Compare PK parameters following a single dose between the two treatment groups following principles of bio-equivalence testing (tmax) | Time period including days 1 to 14 after first infusion in study
  Compare PK parameters following a single dose between the two treatment groups calculating tmax (time to reach maximum serum concentration)
Compare PK parameters following a single dose between the two treatment groups following principles of bio-equivalence testing (t1/2) | Time period including days 1 to 14 after first infusion in study
  Compare PK parameters following a single dose between the two treatment groups calculating t1/2 (apparent terminal half-life)
Compare PK parameters following a single dose between the two treatment groups following principles of bio-equivalence testing (λZ) | Time period including days 1 to 14 after first infusion in study
  Compare PK parameters following a single dose between the two treatment groups calculating λZ (apparent terminal elimination rate constant determined by log-linear regression analysis)
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on occurrence of adverse events | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on occurrence of adverse events
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on blood pressure | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on blood pressure
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on pulse | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on pulse
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on body temperature | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on body temperature
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on respiratory rate | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on respiratory rate
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter hematocrit | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter hematocrit via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter hemoglobin | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter hemoglobin via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter white blood cells | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter white blood cells via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter platelet count | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hematological parameter platelet count via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hepatic parameter alanine aminotransferase | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hepatic parameter alanine aminotransferase via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hepatic parameter aspartate aminotransferase | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring hepatic parameter aspartate aminotransferase via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring renal parameter creatinine | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring renal parameter creatinine via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring renal parameter Blood Urea Nitrogen (BUN) | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on monitoring renal parameter Blood Urea Nitrogen (BUN) via lab test
Evaluate descriptively the safety and tolerability of OctaAlpha1 based on viral safety (HAV, HBV, HCV, HIV-1/2, HN, and parvovirus B19) | 26 weeks
  Evaluate descriptively the safety and tolerability of OctaAlpha1 based on viral safety (HAV, HBV, HCV, HIV-1/2, HN, and parvovirus B19)
Trough Levels of A1PI | 26 weeks
  Investigate descriptively the trough levels of A1PI and anti-NE capacity of OctaAlpha1 compared to Glassia®
Pharmacodynamics of OctaAlpha1 measuring Pulmonary function tests | 26 weeks
  Investigate the pharmacodynamics of OctaAlpha1 measuring Pulmonary function tests (done according to the American Thoracic Society/European Respiratory Society Taskforce Standardisation of Lung Function Testing guideline)
Investigate the pharmacodynamics of OctaAlpha1 measuring Induced sputum test measuring the amount of functional and total A1PI in the airway lining fluid of the lung. | 26 weeks
  Investigate the pharmacodynamics of OctaAlpha1 measuring Induced sputum test measuring the amount of functional and total A1PI in the airway lining fluid of the lung.
Investigate the pharmacodynamics of OctaAlpha1 measuring Induced sputum test measuring the amount of functional and total LTB4 in the airway lining fluid of the lung. | 26 weeks
  Investigate the pharmacodynamics of OctaAlpha1 measuring Induced sputum test measuring the amount of functional and total LTB4 in the airway lining fluid of the lung.
Investigate the pharmacodynamics of OctaAlpha1 measuring antibodies to A1PI using normal ranges of the central laboratory | 26 weeks
  Investigate the pharmacodynamics of OctaAlpha1 measuring antibodies to A1PI using normal ranges of the central laboratory
Determine PK parameters of the A1PI serum concentration versus time curve following a single dose of OctaAlpha1 | 26 weeks
  Determine PK parameters of the A1PI serum concentration versus time curve following a single dose of OctaAlpha1

IPD SHARING:
Plan to Share IPD: Undecided